CLINICAL TRIAL: NCT03946202
Title: Randomised Phase II Trial Testing Efficacy of Intra-tumoural Hydrogen Peroxide as a Radiation Sensitiser in Patients With Locally Advanced/Recurrent Breast Cancer
Brief Title: KORTUC Phase II - Intra-tumoural Radiation Sensitizer in Patients With Locally Advanced/Recurrent Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Kortuc, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR5119; 2019-001709-25 (EudraCT Number)
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Hydrogen Peroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy + radiation sensitiser (Experimental): Patients randomised to the test group will receive standard radiotherapy for breast cancer + a radiation sensitiser
  Interventions: Drug: Hydrogen Peroxide
- Radiotherapy alone (No Intervention): Patients randomised to the control group will receive standard radiotherapy for breast cancer alone

INTERVENTIONS:
Drug: Hydrogen Peroxide — Hydrogen Peroxide
  Arms: Radiotherapy + radiation sensitiser

SUMMARY:
This is a study aimed at testing a commonly available and inexpensive chemical (hydrogen peroxide) for efficacy in sensitising large cancerous lumps in the breast to a standard course of radiotherapy in patients with locally advanced or recurrent breast cancer. Laboratory research and initial clinical trials in Japan suggest that 4 to 6 injections of a radiation sensitiser ('KORTUC') based on very dilute (0.5%) hydrogen peroxide injected into cancers under local anaesthetic twice a week during radiotherapy greatly increases the effectiveness of standard doses of radiotherapy alone. The side effects are limited to mild/moderate discomfort at the injection site for up to 24 hours reported by Japanese breast cancer patients in whom this treatment has been tested. Complete tumour shrinkage in 70/71 (98%) primary breast cancers up to 5 cm diameter have been reported by Japanese collaborators.

DETAILED DESCRIPTION:
Aim: To test a slow release gel containing a commonly available and inexpensive chemical (hydrogen peroxide) for safety and activity in sensitizing large cancerous lumps in the breast or armpit to a standard 3-week course of radiotherapy in patients with locally advanced or recurrent breast cancer.

Background: Laboratory research and initial clinical trials conducted in Japan raises the possibility that a simple and inexpensive treatment based on a very dilute (0.5%) hydrogen peroxide injected into cancers under local anaesthetic greatly increases the effectiveness of standard doses of radiotherapy. The side effects appear to be limited to mild/moderate discomfort at the injection site for up to 24 hours in one-third of patients. Rapid, complete and durable tumour disappearance has been reported in 49/55 bulky breast cancers in Japanese women treated using this approach, a response that is at least 3 times the success rate of radiotherapy alone in our own patients and in a contemporary Japanese control population. The inventor, Prof Ogawa of Kochi University, has approached the investigators to lead the further clinical evaluation and commercial development, starting with the proposed early phase trials testing safety and anti-cancer activity described below.

Design and methods: After numbing the skin with local anaesthetic, a specialist doctor (radiologist) or trained radiographer will use ultrasound to guide the injection of a small volume of dilute (0.5%) hydrogen peroxide solution into the tumour twice a week during 3 weeks of standard radiotherapy. The drug is suspended in a natural gel (1% sodium hyaluronate, licensed for treating stiff knee joints) that ensures its slow release over 48 hours. The injection procedure lasts for 10-15 minutes altogether. Tiny oxygen bubbles are released from the hydrogen peroxide which help the radiologist guide the injection of drug to the proper places under the skin. We have recently completed a safety study confirming the mildness of side effects in 12 patients, and we now wish to test activity against cancer in a randomised controlled trial in 184 patients. Patients participating in Phase II will either have standard radiotherapy or the same radiotherapy plus the drug under test. Neither the patient nor the doctor will choose who has which treatment, which is allocated randomly.

Patient and public involvement: Independent Cancer Patient Voice, a patient advocate group in the field of cancer, is collaborating with the investigators on the research plan, commenting and advising on the content and clarity of the written proposal. This group plays a prominent role in promoting UK clinical research, being represented on the Trial Management Groups of several national randomised cancer clinical trials.

Dissemination: The results of this study will be presented at scientific meetings and at meetings of the patient advocate group in order to judge if the results for safety and activity are promising enough to justify taking the research further.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years and over
* Primary locally advanced breast cancer, or locally recurrent breast cancer with/without metastases (metastases, if present, should be stable or oligometastatic)
* Radical/high dose palliative radiotherapy required for lifetime control of local morbidities
* Patient physically and mentally fit for radical/high dose palliative radiotherapy
* Target tumour accessible for intra-tumoural injection
* Patient suitable/compliant with MR protocol
* At least one tumour diameter ≥30 mm and ≤150 mm measurable by ultrasound or MR imaging
* Patients with predicted life expectancy of 12 months or more
* Negative pregnancy test before start of radiotherapy in women of child bearing potential and an ability/willingness to protect against pregnancy from consent and for 3 months post-radiotherapy
* Patient offers written informed consent

Exclusion Criteria:

* Prior radiotherapy to the target area
* Maximum diameter of target tumour <30 mm or >150mm measurable by ultrasound or MR
* Anatomical location and/or extent of disease difficult to access for safe intra-tumoural drug injections, for example by virtue of contiguous major blood vessels and/or brachial plexus
* Concomitant chemotherapy or biological therapy except Herceptin, Pertuzumab and Denosumab (all endocrine therapies and bisphosphonates are allowed concomitantly; other cytotoxics and biological therapies apart from those mentioned above should be stopped 3 weeks prior to RT)
* Pregnancy or nursing
* Hypersensitivity to any of the KORTUC ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Complete tumour response based on best response assessed by contrast enhanced MRI according to criteria outlined in Section 3.2.1 of the trial protocol, performed up to and including 12 months post radiotherapy | Up to and including 12 months post radiotherapy

SECONDARY OUTCOMES:
Overall survival at 6, 12 and 24 months | 6, 12 and 24 months post radiotherapy
Loco-regional progression-free survival and distant recurrence at 6, 12 and 24 months | 12 and 24 months post radiotherapy
Proportion of patients with either complete response on MRI up to and including 12 months or pathological complete response following tumour resection before 12 months | Up to and including 12 months post radiotherapy
Proportion of patients with partial response and stable disease | 12 and 24 months post radiotherapy
Planned/unplanned tumour excision and pathological response recorded at post-RT follow-up visits | During 24-month follow up period
Adverse events (assessed by NCI CTCAE v5.0) | Up to 90 days post radiotherapy
Compliance with KORTUC injections prior to radiotherapy | During radiotherapy, an average of 3 weeks
Pain at target tumour site following KORTUC injections (10-point scale) | During radiotherapy, an average of 3 weeks
Proportion of patients withdrawing from study due to pain from intratumoural injections recorded at 2-week post-RT visit | During radiotherapy, an average of 3 weeks
Patient-reported quality of life questionnaires (EORTC QLQ-C30 and BR23) | During 24-month follow up period
Resource use and health-related quality of life (EQ-5D-5L) for health economics analysis | During 24-month follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Navita Somaiah, Principal Investigator — The Institute of Cancer Research & The Royal Marsden NHS Foundation Trust
Locations (9):
- India (3):
  - Regional Cancer Centre (RCC), Trivandrum, Kerala
  - Christian Medical Centre, Vellore, Tamil Nadu
  - Tata Medical Centre, Kolkata, West Bengal
- United Kingdom (6):
  - Royal Cornwall Hospitals NHS Trust, Truro, Cornwall
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - The Christie NHS Foundation Trust, Manchester
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Undecided